CLINICAL TRIAL: NCT03990428
Title: A Study to Identify the Supportive Care Needs of Caregivers of Patients With Erdheim-Chester Disease and Other Histiocytic Diseases
Brief Title: Supportive Care Needs of Caregivers of People With Erdheim-Chester Disease and Other Histiocytic Diseases
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-213
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Supportive Care Needs of Caregivers
Keywords: Supportive care; Erdheim-Chester Disease; Other Histiocytic Diseases; 19-213
MeSH Terms: conditions — Erdheim-Chester Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Caregivers of Patients: This is an observational study of informal caregivers (ICs) of patients with Erdheim-Chester Disease (ECD) and other histiocytic diseases. That will collect data cross-sectionally, at a single time point. Caregiver-reported data will be completed in the form of online surveys by the participants themselves using the Research Electronic Data Capture Platform [RedCAP] platform.
  Interventions: Behavioral: online surveys

INTERVENTIONS:
Behavioral: online surveys — Survey data about supportive care needs, mood, and the experience of IC's finding meaning and purpose in the caregiving experience.

SUMMARY:
This study is being done to answer the following question: What are the supportive care needs of informal caregivers of people with Erdheim-Chester disease and other histiocytic diseases?

ELIGIBILITY:
Inclusion Criteria:

* Self-identified informal caregiver (family member or friend who provides unpaid support) for a patient with Erdheim-Chester Disease (or LCH, RDD, or JXG for the exploratory aim).
* Proficiency to complete study assessments in English, evaluated at the time of consent.
* Age 18 or over.

Exclusion Criteria:

* Participant unwilling to sign consent.
* Participant unable to complete web-based assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A target sample of 120 ICs of patients with Erdheim-Chester Disease will be enrolled in this study. Additionally, a target sample of 50 ICs of patients with other histiocytic disorders will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Supportive Care Needs of informal caregivers | 3 years
  measured by the McGill Quality of Life in Life Threatening Illness - Family Carer Version (QLLTI-FC)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm